CLINICAL TRIAL: NCT03694639
Title: CT-guided Ganglion Impar Block for Management of Phantom Rectal Pain Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, lecturer of anesthesia, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MansouraU2
Record Dates: First submitted 2018-09-29; First posted 2018-10-03 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Pain, Phantom
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabaline group (No Intervention): where patients received pregabaline 150 mg twice daily.
- Pregabaline plus ganglion impar block group (Active Comparator): where patients received pregabaline 150 mg twice daily plus ganglion impar block using 5 ml bupivacaine 5% with 14 mg/2 ml betamethasone.
  Interventions: Other: ganglion impar block

INTERVENTIONS:
Other: ganglion impar block — CT sections were done in the axial plane 4 mm slice thickness to detect the site of sacrococcygeal disk. After a suitable section was confirmed, two distances were measured, one from patient's spine to the proper site of entry and the other from the site of entry to the target point.22 gauge spinal needle 12 cm was introduced until reach anterior to sacrococcygeal disk. When the needle tip location was ideal, 2 ml lidocaine mixed with1ml of radiopaque dye was injected. CT sagittal section was done to verify the retroperitoneal distribution of the dye. After good contrast spread confirmation, 5 ml bupivacaine 5% with 14 mg/2 ml betamethasone was injected
  Arms: Pregabaline plus ganglion impar block group

SUMMARY:
Background:Patients underwent abdominoperineal resection with colostomy may suffered from phantom rectum pain syndrome in the perineal area.In this study, the investigators evaluate the combination between ganglion impar block to pregabaline in the treatment of phantom rectal pain syndrome.

Method: Forty patients were randomly allocated into 2 groups: Group A (n=20) where patients received pregabaline 150 mg twice daily. Group B (n=20) where patients received pregabaline 150 mg twice daily plus ganglion impar block using 5 ml bupivacaine 5% with 14 mg/2 ml betamethasone.

DETAILED DESCRIPTION:
Introduction:

Phantom pain syndromes are mostly recorded after amputation of limbs, but it may affect any part of the body (visceral or somatic) has sensory perception following its removal as breast, teeth or rectum.

Patients underwent abdominoperineal resection with colostomy may suffered from phantom rectum pain syndrome in the perineal area characterized as pins, needles, stinging, and burning occurring mostly in sitting positions.

phantom rectum pain syndrome is rarely reported and it is varies from individual to individual. The presence of preoperative rectal pain has a good correlation for the development of postoperative phantom pain.

The pathophysiological mechanisms of phantom phenomena is still unknown but it is neuropathic in nature and believed that it is initiated by changes arising at the peripheral, spinal and supraspinal level leading to central reorganization in additional to the psychogenic factor.

Ganglion impar is a sympathetic ganglion used to manage acute or chronic perineal pain, situated directly in front of the coccyx around the sacrococcygeal joint and behind the rectum in the retroperitoneal space. It can be reached by any guidance as fluoroscopy, computerized tomography, or ultrasound.

Ganglion impar can be done by using multiple methods such as of local anesthetics with steroids or neurolysis by phenol, alcohol and radiofrequency.

The proposal of this study: Is to find the efficacy of the ganglion impar block in patients suffering from phantom rectal pain syndrome after abdominoperineal surgery for rectal cancer with colostomy.

Aim of the work:

To evaluate the combination between ganglion impar block to pregabaline in the treatment of phantom rectal pain syndrome.

Hypothesis:

Management of phantom rectal pain syndrome is a challenging issue needing more appropriate method to reach the best result.

Recharge Gap:

there is a no researches discuss this issue and how to manage it in best way.

Patients and methods:

Study design and participants This randomized pilot controlled study was conducted in pain clinic, Oncology Hospital, Mansoura University during the period from June 2018 till December 2018. The study was accepted by the institutional research board(R.18.09.288 ) . Written informed consents were obtained from forty patients aged from 18 to 70 years of either sex complained from phantom rectal pain syndrome after abdominoperineal surgery for rectal cancer with colostomy.

Patient exclusion criteria include: those who refused to share, evidence of local infection at the puncture site, allergy to drugs used, patients with bleeding tendency or coagulopathy, renal or hepatic failure, cardiac patients, bony abnormality and local malignant recurrence or lower vertebral metastasis.

Routine investigations as complete blood count, coagulation profile (partial thromboplastin time (PTT), prothrombin activity and international normalized ratio (INR)), liver and renal function tests were done prior to procedure. All patients were learned and assessed by numerical rating scale (NRS) for the intensity of pain (If no pain the score was equal zero, if it is worst pain imaginable the score was equal 10).

Sample size:

Internal pilot sample size was estimated on 8 patients during the following period using G-power analysis , assuming α (type I error)=0.05 and β (type II error)= 0.2 (power= 80%) calculate a total sample size of 40.

Patients were randomly allocated into 2 groups:

Group A (n=20) where patients received pregabaline 150 mg twice daily. Group B (n=20) where patients received pregabaline 150 mg twice daily plus ganglion impar block using 5 ml bupivacaine 5% with 14 mg/2 ml betamethasone.

Technique:

Patients were placed in prone position with a cushion under their lower abdomen. CT sections were done in the axial plane 4 mm slice thickness to detect the site of sacrococcygeal disk. After a suitable section was confirmed, two distances were measured, one from patient's spine to the proper site of entry and the other from the site of entry to the target point. Also the angle of needle entrance was calculated. The skin was marked and cleaned with an aseptic solution then anesthetized by 2 ml lidocaine 2%. 22 gauge spinal needle 12 cm was introduced until reach anterior to sacrococcygeal disk. When the needle tip location was ideal, 2 ml lidocaine mixed with1ml of radiopaque dye was injected. CT sagittal section was done to verify the retroperitoneal distribution of the dye. After good contrast spread confirmation, 5 ml bupivacaine 5% with 14 mg/2 ml betamethasone was injected. The patients were observed for one hour after block to note any complication and were discharged at the same day.

ELIGIBILITY:
Inclusion Criteria:

* complained from phantom rectal pain syndrome after abdominoperineal surgery for rectal cancer with colostomy.

Exclusion Criteria:

* those who refused to share
* evidence of local infection at the puncture site
* allergy to drugs used
* patients with bleeding tendency or coagulopathy, renal or hepatic failure, cardiac patients,
* bony abnormality and local malignant recurrence or lower vertebral metastasis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-29 (Estimated)

PRIMARY OUTCOMES:
numerical rating scale | two months
  from 0 to 10 as 0 no pain and 10 the worst pain
Participant satisfaction reporting scale (PSRS) | two months
  it is 5 item self questionnaire1. How well was your pain problem explained to you during treatment?2. Did you agree with the types of treatments and recommendations that you received? 3. How satisfied were you with the care that you received in the Spine Care Center/ Anesthesiology Clinic? 4. Rate your overall improvement since starting treatment: 5. Rate your level of satisfaction with your improvement since starting treatment.

SECONDARY OUTCOMES:
Number of participants with post block complication | 2 hours
  as hematoma, hypotension, neurological defect
success rate of block | one week
  percentage of patients who have numerical rating scale < 4 after one week from block
Pain Anxiety symptoms scale (PASS). | one week
  from 0 to 6 points as 0 = never and 5= always

CONTACTS AND LOCATIONS:
Locations (1):
- Yahay wahba, Al Mansurah, Egypt